CLINICAL TRIAL: NCT05124717
Title: An Open, Comparative, Randomized, Crossover Bioequivalence Study of Single Doses of Metformin, Prolonged-release Tablets 500 mg (JSC Farmak, Ukraine) vs Glucophage® XR 500 mg in Healthy, Adult Male and Female Subjects Under Fed Conditions.
Brief Title: Fed Bioequivalence Study of 2 Metformin 500 mg Prolongued Release Tablets in 28 Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/MTF/FD-500
Record Dates: First submitted 2021-11-09; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Metformin 500 mg Prolonged Release Tablets; Prolonged Release Tablets; oral dosage form; Metformin
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Test Product Metformin, prolonged-release tablets 500 mg (JSC Farmak, Ukraine)
  Interventions: Drug: Metformin, prolonged-release tablets 500 mg (JSC Farmak, Ukraine)
- Treatment B (Active Comparator): Reference Product Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK)
  Interventions: Drug: Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK)

INTERVENTIONS:
Drug: Metformin, prolonged-release tablets 500 mg (JSC Farmak, Ukraine) — One tablet of the Test product was administered orally with 240 mL of water.
  Other Names: Diaformin® SR 500mg tablets (JSC Farmak, Ukraine); Diabufor® XR 500mg tablets (JSC Farmak, Ukraine)
  Arms: Treatment A
Drug: Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK) — One tablet of the Reference product was administered orallyn with 240 mL of water.
  Other Names: Glucophage® XR 500 mg
  Arms: Treatment B

SUMMARY:
The objective of the study is to compare the bioavailability of the Test and Reference products both containing Metformin 500 mg prolonged release tablets (MFM) in healthy male and female volunteers under fed conditions and to assess the bioequivalence of these products based on confidence acceptance intervals of 80.00% to 125.00% for AUC(o-t)and Cmax of MFM as primary endpoints.

DETAILED DESCRIPTION:
An Open, Comparative, Randomized, Crossover Clinical Trial to Evaluate the Bioequivalence of Single Doses of Test Product Metformin, prolonged-release tablets 500 mg (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK) in Healthy, Adult Male and Female Subjects Under Fed Conditions Single oral dose of Glucophage® XR 500 mg prolonged release tablets of Reference product or Metformin, prolonged-release tablets 500 mg of Test product will be administered to volunteers under fed conditions in the morning of Day 1 of each Study Period.

Pharmacokinetic parameters of MFM were calculated from plasma concentrations determined by validated HPLC/MS/MS method.

Pharmacokinetic parameters of the Test and Reference tablets were compared.

During each period 21 samples were taken: prior to dosing (-1.0) and 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, 10.0, 12.0, 16.0, 24.0, 32.0 and 36.0 hours after IMP administration in each study period.

The study consists of two study periods with a washout period of at least 7 days between doses.

Adverse events and clinically significant deviations from laboratory tests, physical examinations and vital signs were reported for the evaluation of safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant and no breast-feeding females (must have a negative pregnancy test result prior to dosing). Caucasian race.
* Non-smoker or past-smoker (who has stopped smoking at least 6 months before the first dosing).
* Body Mass Index (BMI) 18.5 to 30.0 kg/m2, inclusive and body weight between 50 kg and 100 kg(on the day of screening).
* Subject was available for the whole study and has provided his/her written informed consent.
* Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead electrocardiogram (ECG). Minor deviations outside the reference ranges were acceptable, if were deemed not clinically significant by the Investigator.
* Subjects in good health and with glucose between 3.3 mmol/L-5.5 mmol/l at screening, as determined by screening clinical laboratory evaluations. Minor deviations outside the reference ranges were acceptable, if were deemed not clinically significant by the Investigator.
* Acceptance of use of contraceptive measures during the whole study by both female and male subjects.

Exclusion Criteria:

* Known cardiovascular disease, history of hypotension.
* Factors in the subject's history that may predispose to ketoacidosis (including pancreatic insulin deficiency, history of pancreatitis, caloric restriction disoroders, restricted food intake, alcohol abuse)
* Gastrointestinal, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics.
* Previous liver disease or elevations in serum transaminases alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥1.0 upper limit of normal (ULN) at the screening (for women 0-0.52 µmol/L and for men 0-0.68 µmol/L).
* Acute or chronic diseases and/or clinical finding which may interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the Investigational Medicinal Product (IMP).
* History of kidney disease and with impaired renal function.
* History of severe allergy or allergic reactions to the study IMP, its excipients or related drugs.
* Clinically significant illness within 28 days before the first dosing, including major surgery.
* Any significant clinical abnormality including Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and / or (human immunodeficiency virus) HIV. (On screening)
* Positive result of blood pregnancy test at screening or positive urine pregnancy test at check-in or breast-feeding or lack of results of pregnancy test.
* Positive results of drugs of abuse in urine at screening and at check-in.
* Positive result of alcohol breath test at screening and at check-in.
* Positive result of urine cotinine test at screening.
* Serious mental disease and/or inability to cooperate with clinical team.
* Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 90-140 mmHg for systolic blood pressure (BP) and/or 60-90 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
* Body ear temperature is out of the range of 35.7-37.6°C at screening.
* Orthostatic hypotension during the screening procedure.
* Drug, alcohol (of ≥40 g per day pure ethanol), solvents or caffeine abuse.
* Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 90 days before the first dosing.
* Use of any prescription medication for a period of 28 days before the first dosing.
* Use of any OTC (over-the-counter) medication including vitamins, herbal medications and food supplements less than 14 days before the first dosing.
* Getting a tattoo, body piercing or any cosmetic treatment involving skin piercing within 90 days before the screening unless evaluated by Investigator as non-significant for inclusion in the study.
* Donation or loss of at least 500 mL of blood within 90 days or donation of plasma or platelets within 14 days before the first dosing.
* Anaemia, haemoglobin below 120 g/L for women and 130 g/L for men at screening.
* Less than 30 days between exit procedure in previous study and the first dosing in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | up to 36 hours post-administration
  area under the plasma drug concentration versus time curve
Cmax | up to 36 hours post-administration
  maximum plasma concentration observed

SECONDARY OUTCOMES:
AUC(0-∞) | up to 36 hours post-administration
  area under the plasma drug concentration versus time curve from time zero to infinity
AUC(0-12h) | from time zero to time 12 hours after dosing.
  the area under the plasma drug concentration versus time curve calculated from time zero to time 12 hours after dosing
AUC(12h-t) | 12 hours after dosing up to 36 hours post-administration
  the area under the plasma drug concentration versus time curve calculated from time 12 hours after dosing to time of the last sample above LLOQ.
AUC(0-24h) | from time zero to time 24 hours after dosing.
  the area under the plasma drug concentration versus time curve calculated from time zero to time 24 hours after dosing.
tmax | up to 36 hours post-administration
  the time of the maximum plasma drug concentration.
λz | up to 36 hours post-administration
  apparent first-order elimination
AUCres | up to 36 hours post-administration
  Residual area

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- QUINTA-ANALYTICA s.r.o., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No